CLINICAL TRIAL: NCT03862586
Title: Effect of N-Acetyl Cysteine on Expression of HOXA Cluster Genes in Endometrium of Women With Recurrent Implantation Failure (RIF) During Implantation Window: a Double-blinded Randomized Research
Brief Title: NAC Effect on Hox Genes Expressions in RIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Royan-Genetics
Record Dates: First submitted 2018-12-23; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Female Infertility
Keywords: Implantation; Recurrent implantation failure; N-acetyl cysteine; HOXA cluster genes; Window of implantation
MeSH Terms: conditions — Infertility, Female | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetyl cysteine (Experimental): Twenty two infertile women with the onset of endometrial preparation for evaluating genes expression, received 1200 mg of oral N-acetyl cysteine for at-least six weeks before starting ovarian stimulation
  Interventions: Drug: N-acetyl cysteine
- Placebos (Placebo Comparator): Eighteen infertile women with the onset of endometrial preparation for evaluating genes expression, received placebo effervescent tablet for at-least six weeks before starting ovarian stimulation
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: N-acetyl cysteine
  Other Names: NAC
  Arms: N-acetyl cysteine
Drug: Placebos
  Other Names: Placebo effervescent tablet
  Arms: Placebos

SUMMARY:
Comparison of the group treated with NAC-supplementation and placebo- administered groups showed elevations in HOXA cluster genes (all members) expression level in endometrium of women with RIF.

DETAILED DESCRIPTION:
Despite significant developments in assistant reproductive technology (ART) that have overcome many underlying causes of infertility, pregnancy success rates remain relatively low, mainly due to implantation failure. Embryo quality and endometrial receptivity are two significant factors that believed to be the key points in implantation. Since recent studies that showed high expression of some HOXA genes affects on successful implantation rate, thus we examined the expression of HOXA genes in NAC supplementation during window of implantation (WOI) in women with (RIF). Also the effect of NAC on the improvement of implantation in RIF patients was investigated. Forty unfertile women with a diagnosis of RIF, referred to Royan Institute were included in the study. The study was of the type a single center, double blinded, placebo controlled, randomized trial. Expression of HOXA genes were assessed on the day of WOI (using Real Time PCR) biopsies from endometrium. Subjects randomly assigned to receive either NAC (A) or placebo (B) with both effervescent tablets having similar color, size and appearance. The patients were randomly categorized in two groups (A/B) to receive NAC 1200 mg/day or placebo, for at-least 6 weeks before starting ovarian stimulation. Pipelled-based biopsy from endometrium was done on specific day (19-21) of their cycle. Then patients were undergone ovarian stimulation (using NAC) ended to IVF treatment. RNA extraction and cDNA synthesis were performed from endometrium samples and then we evaluated expressions levels by Real-time PCR. Then we analyzed our data by independent Sample T-test and Mann-whitney U Test.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 40 years old
2. At least two IVF failure
3. BMI in the normal range

Exclusion Criteria:

1. Irregular menstrual cycle
2. Taking hormonal drugs except thyroid medication
3. Abnormal karyotype or chromosomal disorders
4. Coagulation problems.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Expression of HOXA in endometrium | approximately 20 days after the first day of menstruation (each day is 28 days)
  mRNA expression by quantitative PCR for homeo box A

SECONDARY OUTCOMES:
Positive pregnancy test | 16 days after embryo transfer
  Measurement of quantitative serum β-hCG
Endometrium thickness | approximately 20 day after the first day of menstruation (each day is 28 days)
  Endometrium thickness

CONTACTS AND LOCATIONS:
Overall Officials: Parvaneh Afsharian, PhD, Study Director — Royan Institute; Ashraf Moini, MD, Study Chair — Royan Institute; Seyed Mehdi Kalantar, PhD, Study Chair — Shahid Sadoughi University of Medical Sciences; Maryam Shahhoseini, PhD, Study Director — Royan Institute; Vida Mokhtari, MSc, Principal Investigator — Royan Institute